CLINICAL TRIAL: NCT01380405
Title: Effectiveness of an Educational Intervention for Managing Inhalers in Chronic Obstructive Pulmonary Disease (COPD) Patients in Primary Care: A Randomized Clinical Trial
Brief Title: Educational Intervention for Managing Inhalers in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: MurciaSalud (Other Government); Public Health Service, Murcia (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRISA II. EPOC-Inhaladores
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inhalators; Education; Primary care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- without health education (No Intervention): the normal practices without specific intervention
- individual health education (Experimental): The study intervention is an individual education in the correct use of inhalers and it will be carried out in so-called "inhalation workshops". The room in which the inhalation workshop will be located has to meet the necessary comfort conditions for the patient to feel relaxed and be able to carry out learning. The lesson included inhalation devices, explanatory leaflets
  Interventions: Behavioral: education intervention
- health education group (Experimental): The study intervention is education in group in the correct use of inhalers and it will be carried out in so-called "inhalation workshops". The room in which the inhalation workshop will be located has to meet the necessary comfort conditions for the patient to feel relaxed and be able to carry out learning. In addition to the necessary furniture and teaching material that will be required (slide projector, over-head-projector, projection screen, video, etc.), the physical space given over to this purpose should consist of an area in which material can be left which will be used to complete the teaching and patient information (inhalation devices, explanatory leaflets, small monographs, slides, etc.).
  Interventions: Behavioral: education intervention

INTERVENTIONS:
Behavioral: education intervention — Individual or collective education interventions about the correct use of inhalers.
  session in the management of inhalers in the collective or individual programmed.
  Session individual: 2 session. 15 min for session. Session collective: 2 session. 30-40 min for session. Maximum 4 persons.
  Arms: health education group; individual health education

SUMMARY:
Given the importance of the correct use of inhalers by patients with Chronic Obstructive Pulmonary Disease (COPD) for the appropriate treatment of the disease, the self-care programme which will be assessed will consist of an educational intervention on the correct use of inhalers.

For this aim, we have designed this study to assess the influence of both individualized and collective self care programmes about the correct use of inhalers improves the functional state of patients with COPD compared to when there is no educational intervention.

DETAILED DESCRIPTION:
One of the key aspects for treating COPD is therapy with inhalation devices. Regarding the correct use of these devices, the international evidence showing that inhalers are not properly used, and in Spain, to the point that the inhaled therapy will fail if it is not accompanied by health education.

More recent studies touch upon the importance of nurses, physicians and other medical staff teaching the correct use of the inhaler. Apart from education, other factors play an important role when it comes to using the inhaler correctly: sex, age, level of education, polymedicated patients who use several kinds of devices, patients who are not aware of their disease and, finally, what is called therapeutic non-fulfillment.

The first report of the effectiveness of a self care programme aimed at the acquisition of self care abilities and behavior change was by Worth. Unfortunately this pilot study was not controlled and only studied a small sample of patients with COPD. There were impressive reductions in the frequency of irritations and house visits by the GP, but no changes in pulmonary function were found.

Several clinical trials have been carried out to evaluate the effectiveness of education programmes and self care in COPD. In the Cochrane revision (up-date 2007), no conclusions could be drawn about the effectiveness of self-control due to the great diversity of variables measured in the few studies published. Based on the antecedents presented, it is evident that COPD is a disease which is difficult to control in daily clinical practice, and that this inadequate control has a significant impact not only on the health of the patient who has this disease, but also on society and the economy.

To improve the control of COPD, the Primary Care physician needs simple and fast intervention to allow him or her to objectively improve the level of control of the disease that these patients have. The objective of self care is to teach patients the necessary aptitudes to carry out specific medical regimes for the treatment of COPD, to guide patients in how to have healthy habits and to lend emotional support to patients to help control their disease

ELIGIBILITY:
The inclusion criteria: A patient diagnosed with COPD undergoing chronic treatment with at least one inhaler in the last year. The criteria of having been prescribed at least 10 prescriptions for an inhaler in the year will be used. Age between 40 to 75 years.

And exclusion criteria: Asthma diagnosis, Serious or terminal illnesses, Limiting osteoarticular disease, Walking disability, Serious mental illnesses: Psychosis, Major depressive disorder, Neurosis, Addictions to drugs/alcohol, Displaced patients (not habitual residents), Pregnancy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To analyze if there is an improvement in the Score of BODE test | 15 days, 30 days, 6 months
  The score is obtained by adding the points together (0-3) for each of the following four variables: distance covered in the 6 minute walking test, forced expiratory volume in the first second in the forced spirometry test, score on the MRC dyspnea test and body mass index

SECONDARY OUTCOMES:
Six minute walking test | 15 days, 30 days, 6 months
Medical Research Council Scale (MRC) to measure the level of dyspnea (Bestall y col). | 15 days, 30 days, 6 months
Number of recurrences | 15 days, 30 days, 6 months
Number of hospitalisations | 15 days, 30 days, 6 months
Visual assessment scales of the use of inhalers | 15 days, 30 days, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: A Lopez-Santiago, MD, Principal Investigator — Consejeria de sanidad y consumo, Direccion general de planificacion, ordenacion sanitaria y farmaceutica e investigacion.
Locations (1):
- Fundación para la Formación e Investigación Sanitarias de la Región de Murcia, Murcia, Murcia, Spain

REFERENCES:
- [Background] Annesi- Maesano I. Epidemiology of chronic obstructive pulmonary disease. In: Siafakas NM, ed. Management of Chronic Obstructive Pulmonary Disease. 2006.
- [Background] Sobradillo V, Miravitlles M, Jimenez CA, Gabriel R, Viejo JL, Masa JF, Fernandez-Fau L, Villasante C. [Epidemiological study of chronic obstructive pulmonary disease in Spain (IBERPOC): prevalence of chronic respiratory symptoms and airflow limitation]. Arch Bronconeumol. 1999 Apr;35(4):159-66. doi: 10.1016/s0300-2896(15)30272-6. Spanish. PMID 10330536
- [Background] Miravitlles M, Soriano JB, Garcia-Rio F, Munoz L, Duran-Tauleria E, Sanchez G, Sobradillo V, Ancochea J. Prevalence of COPD in Spain: impact of undiagnosed COPD on quality of life and daily life activities. Thorax. 2009 Oct;64(10):863-8. doi: 10.1136/thx.2009.115725. Epub 2009 Jun 23. PMID 19553233
- [Background] Masa JF, Sobradillo V, Villasante C, Jimenez-Ruiz CA, Fernandez-Fau L, Viejo JL, Miravitlles M. [Costs of chronic obstructive pulmonary disease in Spain. Estimation from a population-based study]. Arch Bronconeumol. 2004 Feb;40(2):72-9. doi: 10.1016/s1579-2129(06)60198-5. Spanish. PMID 14746730
- [Background] Instituto Nacional de Estadística INE. Encuesta Nacional de Salud 2006.
- [Background] Peces-Barba G, Barbera JA, Agusti A, Casanova C, Casas A, Izquierdo JL, Jardim J, Lopez Varela V, Monso E, Montemayor T, Viejo JL. [Diagnosis and management of chronic obstructive pulmonary disease: joint guidelines of the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR) and the Latin American Thoracic Society (ALAT)]. Arch Bronconeumol. 2008 May;44(5):271-81. No abstract available. Spanish. PMID 18448019
- [Background] Haupt D, Krigsman K, Nilsson JL. Medication persistence among patients with asthma/COPD drugs. Pharm World Sci. 2008 Oct;30(5):509-14. doi: 10.1007/s11096-008-9197-4. Epub 2008 Feb 5. PMID 18247154
- [Background] Jung E, Pickard AS, Salmon JW, Bartle B, Lee TA. Medication adherence and persistence in the last year of life in COPD patients. Respir Med. 2009 Apr;103(4):525-34. doi: 10.1016/j.rmed.2008.11.004. Epub 2009 Jan 12. PMID 19136240
- [Background] Burgos F. [Inhalation therapy without instruction: failure foreseen]. Arch Bronconeumol. 2002 Jul;38(7):297-9. doi: 10.1016/s0300-2896(02)75221-6. No abstract available. Spanish. PMID 12199927
- [Background] Flor Escriche X, Rodriguez Mas M, Gallego Alvarez L, Alvarez Luque I, Juvanteny Gorgals J, Fraga Martinez MM, Sanchez Pinacho L. [Do our asthma patients still use inhalers incorrectly?]. Aten Primaria. 2003 Sep 30;32(5):269-74. doi: 10.1016/s0212-6567(03)79273-7. Spanish. PMID 14519287
- [Background] Bourbeau J, Julien M, Maltais F, Rouleau M, Beaupre A, Begin R, Renzi P, Nault D, Borycki E, Schwartzman K, Singh R, Collet JP; Chronic Obstructive Pulmonary Disease axis of the Respiratory Network Fonds de la Recherche en Sante du Quebec. Reduction of hospital utilization in patients with chronic obstructive pulmonary disease: a disease-specific self-management intervention. Arch Intern Med. 2003 Mar 10;163(5):585-91. doi: 10.1001/archinte.163.5.585. PMID 12622605
- [Background] Worth H. Self management in COPD: one step beyond? Patient Educ Couns. 1997 Dec;32(1 Suppl):S105-9. doi: 10.1016/s0738-3991(97)00102-x. PMID 9516766
- [Background] Effing T, Monninkhof EM, van der Valk PD, van der Palen J, van Herwaarden CL, Partidge MR, Walters EH, Zielhuis GA. Self-management education for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD002990. doi: 10.1002/14651858.CD002990.pub2. PMID 17943778
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh?term=inhalators
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh/68011320
- See also: MeSH — http://www.ncbi.nlm.nih.gov/mesh?term=education